CLINICAL TRIAL: NCT04016480
Title: High Flow Oxygen Therapy Through Nasal Cannula in Patients With Acute Respiratory Failure During Bronchoscopy for Bronchoalveolar Lavage
Brief Title: HFNC During Bronchoscopy for Bronchoalveolar Lavage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Principal Investigator, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFNC-FBS
Record Dates: First submitted 2019-07-02; First posted 2019-07-11 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Acute Respiratory Failure; Bronchoscopy; Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (Active Comparator): High Flow Nasal cannula is a system to deliver heated and humidified oxygen with an inspired oxygen fraction between 21 and 100% through large bore nasal cannula. The system delivers a flow up to 60 liters/min.
  Interventions: Device: High Flow Nasal Cannula
- Conventional Oxygen Therapy (Active Comparator): Conventional oxygen therapy will be administered through common nasal cannula with a flow up to 6 Liters per minute
  Interventions: Device: Conventional Oxygen Therapy

INTERVENTIONS:
Device: High Flow Nasal Cannula — High Flow Nasal Cannula will be set at 60 liters per minute of air/oxygen admixture to reach a peripheral oxygen saturation equal or greater than 94%
  Arms: High Flow Nasal Cannula
Device: Conventional Oxygen Therapy — Conventional Oxygen Therapy will be administered through nasal cannula with a oxygen flow set to achieve a peripheral oxygen saturation equal or greater than 94%
  Arms: Conventional Oxygen Therapy

SUMMARY:
The execution of diagnostic-therapeutic investigations by bronchial endoscopy can expose the patient to acute respiratory failure (ARF). In particular, the risk of hypoxemia is greater during broncho-alveolar lavage (BAL). For this reason, oxygen therapy is administered at low or high flows during the course of bronchoscopic procedures, in order to avoid hypoxemia.

Few clinical studies have demonstrated the efficacy and safety of high flow oxygen through nasal cannula (HFNC) during BAL procedures, and no study has evaluated, during bronchial endoscopy, the effects of HFNC on diaphragmatic effort (assessed with ultrasound) and aeration and ventilation of the different lung regions (assessed with electrical impedance tomography).

Therefore, investigators conceived the present randomized controlled study to evaluate possible differences existing during bronchoscopy between oxygen therapy administered with HFNC and conventional (low-flow) oxygen therapy, delivered through nasal cannula.

DETAILED DESCRIPTION:
Patients with Acute Respiratory Failure may sometimes require a bronchial endoscopy for broncho-alveolar lavage (BAL).

During the procedure, hypoxemia may worsen and oxygen may be require to avoid desaturation.

In the recent years, High-Flow through Nasal Cannula (HFNC) has been introduced in the clinical practice. HFNC delivers to the patient heated humidified air-oxygen mixture, with an inspiratory fraction of oxygen (FiO2) ranging from 21 to 100% and a flow up to 60 L/min through a large bore nasal cannula.

HFNC has some potential advantages. First of all, HFNC provides heated (37°C) and humidified (44 mg/L) air-oxygen admixture to the patient, which avoids injuries to ciliary motion, reduces the inflammatory responses associated to dry and cold gases, epithelial cell cilia damage, and airway water loss, and keeps unmodified the water content of the bronchial secretions. Second, HFNC determines a wash out from carbon dioxide of the pharyngeal dead space. Third, HFNC generates small amount (up to 8 cmH2O) of pharyngeal pressure during expiration, which drops to zero during inspiration. Fourth, HFNC guarantees a more stable FiO2, as compared to conventional oxygen therapy. Whenever the inspiratory peak flow of a patient exceeds the flow provided by a Venturi mask, the patient inhaled also part of atmospheric air.

Electrical impedance tomography (EIT) is a noninvasive imaging technique providing instantaneous monitoring of variations in overall lung volume and regional distribution of ventilation, as determined by variations over time in intrathoracic impedance, which is increased by air and reduced by fluids and cells. EIT allows determining changes in end-expiratory lung impedance (EELI), a surrogate estimate of end-expiratory lung volume, assessing global and regional distribution of Vt, and obtaining indexes of spatial distribution of ventilation.

Diaphragm ultrasound is a bedside, radiation free technique to assess the contractility of the diaphragm and the respiratory effort.

In this study investigators aim to evaluate possible differences existing during bronchoscopy between oxygen therapy administered with HFNC and conventional (low-flow) oxygen therapy, delivered through nasal cannula in terms of respiratory effort (as assessed through diaphragm ultrasound), lung aeration and ventilation distribution (as assessed with EIT) and arterial blood gases.

ELIGIBILITY:
Inclusion Criteria:

* need for bronchial endoscopy for bronchoalveolar lavage

Exclusion Criteria:

* life-threatening cardiac aritmia or acute miocardical infarction within 6 weeks
* need for invasive or non invasive ventilation
* presence of pneumothorax or pulmonary enphisema or bullae
* recent (within 1 week) thoracic surgery
* presence of chest burns
* presence of tracheostomy
* pregnancy
* nasal or nasopharyngeal diseases
* dementia
* lack of consent or its withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Arterial blood gases at end of the procedure | After 0 minute from the end of the bronchial endoscopy
  Arterial blood will be sample for gas analysis

SECONDARY OUTCOMES:
Respiratory effort at end of the procedure | After 0 minute from the end of the bronchial endoscopy
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Respiratory effort at baseline | After 0 minute from enrollment
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Respiratory effort at the beginning of the bronchoscopy | 5 minutes before the beginning of the bronchial endoscopy, while receiving the assigned treatment
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Respiratory effort after bronchoscopy | After 10 minute from the end of the bronchial endoscopy
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Change of end-expiratory lung impedance (dEELI) from baseline at the beginning of the bronchoscopy | 5 minutes before the beginning of the bronchial endoscopy, while receiving the assigned treatment, compared to baseline
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of end-expiratory lung impedance (dEELI) from baseline at end of the procedure | After 0 minute from the end of the bronchial endoscopy, compared to baseline
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of end-expiratory lung impedance (dEELI) from baseline after bronchoscopy | After 10 minute from the end of the bronchial endoscopy, compared to baseline
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from baseline at the beginning of bronchoscopy | 5 minutes before the beginning of the bronchial endoscopy, while receiving the assigned treatment, compared to baseline
  change from baseline, expressed in percentage, of the tidal volume as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from baseline at end of the procedure | After 0 minute from the end of the bronchial endoscopy, compared to baseline
  change from baseline, expressed in percentage, of the tidal volume as assessed through electrical impedance tomography
Change of tidal volume in percentage (dVt%) from baseline after bronchoscopy | After 10 minute from the end of the bronchial endoscopy, compared to baseline
  change from baseline, expressed in percentage, of the tidal volume as assessed through electrical impedance tomography
Arterial blood gases at baseline | After 0 minute from enrollment
  Arterial blood will be sample for gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, datasets used and analysed during the current study will be available on reasonable request e-mailing the corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared after results publication of indexed journal in english language
Access Criteria: On reasonable request

REFERENCES:
- [Background] Albertini R, Harrel JH, Moser KM. Letter: Hypoxemia during fiberoptic bronchoscopy. Chest. 1974 Jan;65(1):117-8. doi: 10.1378/chest.65.1.117. No abstract available. PMID 4809326
- [Background] Randazzo GP, Wilson AR. Cardiopulmonary changes during flexible fiberoptic bronchoscopy. Respiration. 1976;33(2):143-9. doi: 10.1159/000193727. PMID 935677
- [Background] Pirozynski M, Sliwinski P, Radwan L, Zielinski J. Bronchoalveolar lavage: comparison of three commonly used procedures. Respiration. 1991;58(2):72-6. doi: 10.1159/000195900. PMID 1862254
- [Background] Cuquemelle E, Pham T, Papon JF, Louis B, Danin PE, Brochard L. Heated and humidified high-flow oxygen therapy reduces discomfort during hypoxemic respiratory failure. Respir Care. 2012 Oct;57(10):1571-7. doi: 10.4187/respcare.01681. Epub 2012 Mar 12. PMID 22417569
- [Background] Renda T, Corrado A, Iskandar G, Pelaia G, Abdalla K, Navalesi P. High-flow nasal oxygen therapy in intensive care and anaesthesia. Br J Anaesth. 2018 Jan;120(1):18-27. doi: 10.1016/j.bja.2017.11.010. Epub 2017 Nov 21. PMID 29397127
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Miyagi K, Haranaga S, Higa F, Tateyama M, Fujita J. Implementation of bronchoalveolar lavage using a high-flow nasal cannula in five cases of acute respiratory failure. Respir Investig. 2014 Sep;52(5):310-4. doi: 10.1016/j.resinv.2014.06.006. Epub 2014 Jul 25. PMID 25169847
- [Background] Kim EJ, Jung CY, Kim KC. Effectiveness and Safety of High-Flow Nasal Cannula Oxygen Delivery during Bronchoalveolar Lavage in Acute Respiratory Failure Patients. Tuberc Respir Dis (Seoul). 2018 Oct;81(4):319-329. doi: 10.4046/trd.2017.0122. Epub 2018 Jun 19. PMID 29926546
- [Background] Longhini F, Pisani L, Lungu R, Comellini V, Bruni A, Garofalo E, Laura Vega M, Cammarota G, Nava S, Navalesi P. High-Flow Oxygen Therapy After Noninvasive Ventilation Interruption in Patients Recovering From Hypercapnic Acute Respiratory Failure: A Physiological Crossover Trial. Crit Care Med. 2019 Jun;47(6):e506-e511. doi: 10.1097/CCM.0000000000003740. PMID 30882477
- [Derived] Longhini F, Pelaia C, Garofalo E, Bruni A, Placida R, Iaquinta C, Arrighi E, Perri G, Procopio G, Cancelliere A, Rovida S, Marrazzo G, Pelaia G, Navalesi P. High-flow nasal cannula oxygen therapy for outpatients undergoing flexible bronchoscopy: a randomised controlled trial. Thorax. 2022 Jan;77(1):58-64. doi: 10.1136/thoraxjnl-2021-217116. Epub 2021 Apr 29. PMID 33927023